CLINICAL TRIAL: NCT01311427
Title: Simplified Tai Chi for Reducing Fibromyalgia Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Responsible Party: Kim D. Jones, Associate Professor, Oregon Health & Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIAMS 5R21 AR053506
Record Dates: First submitted 2011-02-09; First posted 2011-03-09 (Estimated); Last update posted 2011-03-09 (Estimated); Status verified 2011-03

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group education (Active Comparator): The control condition received standard group education, which met in small groups two times weekly for 60 minutes over 12 weeks.
  Interventions: Behavioral: Group education
- 8-form Yang-style Tai chi program (Experimental): This arm tested a modified 8-form Yang-style Tai chi program in subjects with fibromyalgia. Participants met in small groups two times weekly for 60 minutes over 12 weeks.
  Interventions: Behavioral: 8-form Yang-style Tai chi

INTERVENTIONS:
Behavioral: 8-form Yang-style Tai chi — This study tested a modified 8-form Yang-style Tai chi program in subjects with fibromyalgia. Participants met in a small group two times weekly for 60 minutes over 12 weeks.
  Arms: 8-form Yang-style Tai chi program
Behavioral: Group education — Standard group education was delivered to participants in a small group format twice weekly for 60 minutes over 12 weeks.
  Arms: Group education

SUMMARY:
Data from two recent Tai chi studies have found that Tai Chi yields symptomatic benefit in patients with fibromyalgia (FM). The purpose of this study is to confirm those findings in a larger randomized, controlled clinical trial in a community-based setting. We also sought to extend this line of inquiry by closely examining Tai chi's effect on physical function, specifically postural stability. Towards these ends, we conducted a single-blind, randomized controlled clinical trial of an FM modified 8-form Yang-style Tai chi program compared to standard education. Subjects in both conditions meet in small groups two times weekly for 60 minutes over 12 weeks.

DETAILED DESCRIPTION:
120 males and females with fibromyalgia were randomized to participate in a modified 8 form Yang-Style Tai Chi program or a standard group education program. Both programs met in a small group format for twice weekly 60 minute sessions lasting for 12 weeks. 99 subjects completed the protocol. Primary outcomes from the Fibromyalgia Impact Questionnaire were assessed at baseline and 12 weeks. Secondary measures included pain intensity and interference, sleep, coping, and fitness tests.

ELIGIBILITY:
Inclusion Criteria:

* Subjects included adults over 40 years of age or older who met 1990 ACR criteria for the classification of FM. Those criteria include pain in three or more body quadrants (above the waist, below the waist, left of midline and right of midline) including axial pain by self-report for a minimum of three consecutive months.
* Additionally at least 11 of 18 muscle/tendon junction tender points were found to be painful via digital palpation of 4kg over 4 seconds by a trained examiner (Wolfe 1990).

Exclusion Criteria:

* Individuals were excluded if they practiced Tai chi within the past 6 months; - were exercising more than 30 minutes, three times weekly for past 3 months;
* could not independently ambulate without assistive devices;
* were unable to attain MD clearance for exercise within past 3 months;
* were unwilling to undergo random assignment; had cognitive impairment based on score >3 Pfeiffer Mental Status;
* had significant depressive symptoms based on a score of >27 on Beck Depression Inventory;
* had BPI pain severity scores less than 3/10, had planned elective surgery during the study period;
* were unwilling to keep all treatments/medications steady throughout the study period;
* were currently enrolled in another study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2006-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire | Assessed following 12 week intervention

SECONDARY OUTCOMES:
Brief Pain Inventory | Assessed following 12 week intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kim D Jones, PhD, Study Chair — Oregon Health and Science University
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States

REFERENCES:
- [Derived] Jones KD, Sherman CA, Mist SD, Carson JW, Bennett RM, Li F. A randomized controlled trial of 8-form Tai chi improves symptoms and functional mobility in fibromyalgia patients. Clin Rheumatol. 2012 Aug;31(8):1205-14. doi: 10.1007/s10067-012-1996-2. Epub 2012 May 13. PMID 22581278